CLINICAL TRIAL: NCT05354375
Title: Clinical Study of PSMA-targeted CAR-T Cells in the Treatment of Castration-resistant Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Collaborators: Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2021-KL172-02
Record Dates: First submitted 2022-04-26; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2021-11

CONDITIONS: Immunotherapy
Keywords: Prostate specific membrane antigen; Castration-resistant Prostate Cancer; CAR-T; Chimeric antigen receptor; T cell
MeSH Terms: interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T cell immunotherapy (Experimental): The registered patients will receive CAR-T cell immunotherapy for the new specific chimeric antigen receptor of PSMA antigen by infusion.
  Interventions: Biological: CAR-T cell immunotherapy

INTERVENTIONS:
Biological: CAR-T cell immunotherapy — This CAR-T cell immunotherapy with a novel specific Chimeric antigen receptor aiming at PSMA.

SUMMARY:
This is an experimental study to evaluate the safety and effectiveness of PSMA-targeted CAR-T cells in the treatment of castration-resistant prostate cancer.

DETAILED DESCRIPTION:
We designed a clinical study and divided the trial into two phases.

Phase 1 (climbing test): 9 patients were randomly divided into 3 groups (n=3). 9 patients were treated with cyclophosphamide at the dose of 60mg/kg/d 8-7 days before CAR-T cell infusion, and fludalabine at the dose of 25mg/m^2/d 6-2 days before CAR-T cell infusion. On Day 0, CAR T cells were injected into patients in group 1, 2 and 3 at the dose of 1*10^8/ person, 1*10^9/ person and 1*10^10/ person, respectively. The infusion time exceeded 15-30min. On day 0-14, IL-2 (75000IU/kg) was injected subcutaneously once a day. From day 15-28, IL-2 (75000IU/kg) was subcutaneously injected into the patients three times a week. The purpose of this study is to assess subjects' MTD (maximum tolerated dose) against CAR T cells.

Phase 2: After determining the appropriate therapeutic dose for patients with prostate cancer, the remaining 11 patients received the same pre-treatment of chemotherapy. Then, the appropriate therapeutic dose of CAR T cells according to the results of phase 1 was infused on Day 0. On day 0-14,IL-2 (75000IU/kg) was given subcutaneously once a day. On day 15-28, IL-2 (75000IU/kg) was given subcutaneously three times a week.

Subjects will collect peripheral blood every four weeks, detect PSA and other related indicators to evaluate the curative effect, safety and survival rate of CAR-T cell transplantation. After 6 months of close follow-up, the subjects will have a quarterly medical history assessment, physical examination and blood test, bone metastasis assessment by bone ECT, prostate and pelvic cavity assessment by prostate MRI, and general information by PET CT if necessary for two years. After this assessment, the subjects will enter an annual telephone follow-up and questionnaire survey for up to five years to assess the long-term health problems of treatment, such as recurrence of malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients aged from 18 to 75 years old;
2. The patients' ECOG score ≤ 2;
3. Prostate cancer patients in castration resistance stage (with or without distant metastasis):

   1. Previous new endocrine therapy is ineffective;
   2. Past treatment with too much citabine or cabatase is ineffective.
4. Have measurable or evaluable lesions;
5. The patients' main tissues and organs function well:

   1. Liver function: ALT/AST < 3 times the upper limit of normal value (ULN);
   2. renal function: creatinine < 220 μ mol/L;
   3. Lung function: indoor oxygen saturation ≥ 95%;
   4. Cardiac function: Left ventricular ejection fraction (LVEF)≥40%
6. Patients or their legal guardians voluntarily participate and sign the informed consent form.

Exclusion Criteria:

1. Infectious diseases (such as HIV, active hepatitis B or C infection, active tuberculosis, etc.);
2. Feasibility evaluation screening proves that the transfection of targeted lymphocytes is less than 10% or the amplification under the co-stimulation of CD3/CD28 is insufficient (< 5 times);
3. The vital signs are abnormal and those who cannot cooperate with the inspectors;
4. Those with mental illness or mental illness who can't cooperate with treatment and curative effect evaluation;
5. Highly allergic constitution or severe allergic history, especially those who are allergic to IL-2;
6. Subjects with systemic infection or local severe infection who need anti-infection treatment;
7. Complicated dysfunction of heart, lung, brain, liver, kidney and other important organs;
8. Patients with other tumors;
9. Doctors think that there are other reasons that can't be included in the treatment.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety Evaluation:Incidence and Severity of Adverse Events | First 1 month after CAR-T cells infusion
  To evaluate the incidence and severity of possible adverse events within one month after targeted PSMA CAR-T infusion, including cytokine release syndrome and on-target toxicity.
Effectiveness Evaluation | 3 months after CAR-T cells infusion
  In order to observe the efficacy of CAR-T cells after infusion, total remission rate (ORR), complete remission (CR), partial remission (PR), disease stability (SD) or progression (PD) will be used for evaluation.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) | 24 months after CAR-T cells infusion
  Progression-free survival (PFS) time
Overall Survival (OS) | 24 months after CAR-T cells infusion
  Overall survival (OS) time

CONTACTS AND LOCATIONS:
Overall Officials: Junnian Zheng, M.D/Ph.D, Study Director — The Affiliated Hospital of Xuzhou Medical University; Hailong Li, M.D/Ph.D, Principal Investigator — The Affiliated Hospital of Xuzhou Medical University; Qing Zhang, Ph.D, Principal Investigator — Xuzhou Medical University
Locations (1):
- Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mohler JL, Antonarakis ES, Armstrong AJ, D'Amico AV, Davis BJ, Dorff T, Eastham JA, Enke CA, Farrington TA, Higano CS, Horwitz EM, Hurwitz M, Ippolito JE, Kane CJ, Kuettel MR, Lang JM, McKenney J, Netto G, Penson DF, Plimack ER, Pow-Sang JM, Pugh TJ, Richey S, Roach M, Rosenfeld S, Schaeffer E, Shabsigh A, Small EJ, Spratt DE, Srinivas S, Tward J, Shead DA, Freedman-Cass DA. Prostate Cancer, Version 2.2019, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2019 May 1;17(5):479-505. doi: 10.6004/jnccn.2019.0023. PMID 31085757
- [Result] Gansler T, Ganz PA, Grant M, Greene FL, Johnstone P, Mahoney M, Newman LA, Oh WK, Thomas CR Jr, Thun MJ, Vickers AJ, Wender RC, Brawley OW. Sixty years of CA: a cancer journal for clinicians. CA Cancer J Clin. 2010 Nov-Dec;60(6):345-50. doi: 10.3322/caac.20088. PMID 21075954
- [Result] Slovin SF. Immunotherapy for castration-resistant prostate cancer: has its time arrived? Expert Opin Biol Ther. 2020 May;20(5):481-487. doi: 10.1080/14712598.2020.1735345. Epub 2020 Mar 5. PMID 32097050
- [Result] Esmaeilzadeh A, Tahmasebi S, Athari SS. Chimeric antigen receptor -T cell therapy: Applications and challenges in treatment of allergy and asthma. Biomed Pharmacother. 2020 Mar;123:109685. doi: 10.1016/j.biopha.2019.109685. Epub 2019 Dec 17. PMID 31862474
- [Result] Zuccolotto G, Fracasso G, Merlo A, Montagner IM, Rondina M, Bobisse S, Figini M, Cingarlini S, Colombatti M, Zanovello P, Rosato A. PSMA-specific CAR-engineered T cells eradicate disseminated prostate cancer in preclinical models. PLoS One. 2014 Oct 3;9(10):e109427. doi: 10.1371/journal.pone.0109427. eCollection 2014. PMID 25279468
- [Result] Minn I, Huss DJ, Ahn HH, Chinn TM, Park A, Jones J, Brummet M, Rowe SP, Sysa-Shah P, Du Y, Levitsky HI, Pomper MG. Imaging CAR T cell therapy with PSMA-targeted positron emission tomography. Sci Adv. 2019 Jul 3;5(7):eaaw5096. doi: 10.1126/sciadv.aaw5096. eCollection 2019 Jul. PMID 31281894
- [Result] Santoro SP, Kim S, Motz GT, Alatzoglou D, Li C, Irving M, Powell DJ Jr, Coukos G. T cells bearing a chimeric antigen receptor against prostate-specific membrane antigen mediate vascular disruption and result in tumor regression. Cancer Immunol Res. 2015 Jan;3(1):68-84. doi: 10.1158/2326-6066.CIR-14-0192. Epub 2014 Oct 30. PMID 25358763
- [Result] Zhang Q, Li H, Yang J, Li L, Zhang B, Li J, Zheng J. Strategies to improve the clinical performance of chimeric antigen receptor-modified T cells for cancer. Curr Gene Ther. 2013 Feb;13(1):65-70. doi: 10.2174/156652313804806570. PMID 23256743
- [Result] Sadelain M, Riviere I, Riddell S. Therapeutic T cell engineering. Nature. 2017 May 24;545(7655):423-431. doi: 10.1038/nature22395. PMID 28541315
- [Result] Xu J, Tian K, Zhang H, Li L, Liu H, Liu J, Zhang Q, Zheng J. Chimeric antigen receptor-T cell therapy for solid tumors require new clinical regimens. Expert Rev Anticancer Ther. 2017 Dec;17(12):1099-1106. doi: 10.1080/14737140.2017.1395285. Epub 2017 Oct 26. PMID 29048935
- [Result] Junghans RP, Ma Q, Rathore R, Gomes EM, Bais AJ, Lo AS, Abedi M, Davies RA, Cabral HJ, Al-Homsi AS, Cohen SI. Phase I Trial of Anti-PSMA Designer CAR-T Cells in Prostate Cancer: Possible Role for Interacting Interleukin 2-T Cell Pharmacodynamics as a Determinant of Clinical Response. Prostate. 2016 Oct;76(14):1257-70. doi: 10.1002/pros.23214. Epub 2016 Jun 21. PMID 27324746